CLINICAL TRIAL: NCT02627677
Title: A Randomized, Open-label Study of Ponatinib Versus Nilotinib in Patients With Chronic Myeloid Leukemia in Chronic Phase Following Resistance to Imatinib
Brief Title: A Study Comparing Ponatinib and Nilotinib in Participants With Chronic Myeloid Leukemia
Acronym: OPTIC-2L
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to operational feasibility and not due to any safety concerns
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP24534-15-303; 2015-001318-92 (EudraCT Number)
Record Dates: First submitted 2015-08-13; First posted 2015-12-11 (Estimated); Results first posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-10

CONDITIONS: Chronic Phase Chronic Myeloid Leukemia
Keywords: CML; CP-CML; Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms by Histologic Type; Neoplasms; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia; Leukemia, Myeloid; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Neoplasms by Histologic Type; Neoplasms; Myeloproliferative Disorders; Bone Marrow Diseases; Hematologic Diseases | interventions — ponatinib; nilotinib; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Ponatinib 30 mg (Experimental): Ponatinib 30 mg, tablets, orally, once daily (QD) until achievement of major molecular response (MMR) up to 12 months. Once MMR was achieved, participants received reduced dose of ponatinib 15 mg orally once daily up to 42 months.
  Interventions: Drug: Ponatinib 30 mg QD
- Cohort B: Ponatinib 15 mg (Experimental): Ponatinib 15 mg, tablets, orally, QD until achievement of MMR up to 12 months. Once MMR was achieved, participants received reduced dose of ponatinib 15 mg orally once daily up to 45 months.
  Interventions: Drug: Ponatinib 15 mg QD
- Cohort C: Nilotinib 400 mg (Active Comparator): Nilotinib 400 mg, tablets, orally, twice daily up to approximately 42 months.
  Interventions: Drug: Nilotinib 400 mg BID

INTERVENTIONS:
Drug: Ponatinib 30 mg QD — Ponatinib 30 mg, taken orally once daily.
  Other Names: Iclusig; AP24534
  Arms: Cohort A: Ponatinib 30 mg
Drug: Ponatinib 15 mg QD — Ponatinib 15 mg, taken orally once daily.
  Other Names: Iclusig; AP24534
  Arms: Cohort B: Ponatinib 15 mg
Drug: Nilotinib 400 mg BID — Nilotinib 400 mg, taken orally twice daily.
  Other Names: Tasigna; AMN107
  Arms: Cohort C: Nilotinib 400 mg

SUMMARY:
The purpose of this study is to compare the efficacy and safety of 2 starting doses of ponatinib compared to nilotinib in participants with imatinib-resistant chronic myeloid leukemia (CML) in chronic phase (CP).

DETAILED DESCRIPTION:
This is a multi-center, randomized study to demonstrate the efficacy and safety of 2 starting doses of ponatinib as a treatment for CP-CML compared to nilotinib. Eligible participants must have chronic phase chronic myeloid leukemia (CP-CML), be resistant to first-line imatinib treatment and have received no other tyrosine kinase inhibitors (TKIs).

ELIGIBILITY:
Inclusion Criteria:

1. Have CP-CML and are resistant to first-line imatinib treatment.
2. Be male or female ≥18 years old.
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Have adequate renal function as defined by the following criterion:

   • Serum creatinine ≤1.5 × upper limit of normal (ULN) for institution.
5. Have adequate hepatic function as defined by all of the following criteria:

   * Total serum bilirubin ≤1.5 × ULN, unless due to Gilbert's syndrome
   * Alanine aminotransferase (ALT) ≤2.5 × ULN or ≤5 × ULN if leukemic infiltration of the liver is present
   * Aspartate aminotransferase (AST) ≤2.5 × ULN or ≤5 × ULN if leukemic infiltration of the liver is present.
6. Have normal pancreatic status as defined by the following criterion:

   * Serum lipase and amylase ≤1.5 × ULN.

Exclusion Criteria:

1. Have previously been treated with any approved or investigational TKIs other than imatinib or treated with imatinib within 14 days prior to receiving study drug.
2. Have previously been treated with any anti-CML therapy other than hydroxyurea, including interferon, cytarabine, immunotherapy, or any cytotoxic chemotherapy, radiotherapy, or investigational therapy.
3. Underwent autologous or allogeneic stem cell transplant.
4. Are in CCyR or MMR.
5. Have clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   * Any history of myocardial infarction (MI), unstable angina, cerebrovascular accident, or transient ischemic attack (TIA)
   * Any history of peripheral vascular infarction, including visceral infarction
   * Any history of a revascularization procedure, including vascular surgery or the placement of a stent
   * History of venous thromboembolism, including deep venous thrombosis, superficial venous thrombosis, or pulmonary embolism, within 6 months prior to enrollment
   * Congestive heart failure (New York Heart Association [NYHA] class III or IV) within 6 months prior to enrollment or left ventricular ejection fraction (LVEF) less than 45% or less than the institutional lower limit of normal (whichever is higher) within 6 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2021-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Cliniques Universitaire Saint-Luc (Site 058), Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 90 investigative sites in Austria, Canada, Czechia, France, Hungary, Italy, Korea, and Russia from 31 December 2015 to 20 January 2021
Pre-assignment Details: Participants with a diagnosis of chronic phase-chronic myeloid leukemia were enrolled and randomised at a ratio of 1:2:1 to receive ponatinib 30 mg and ponatinib 15 mg compared with nilotinib 400 mg.
Groups:
- Cohort A: Ponatinib 30 mg: Ponatinib 30 mg, tablets, orally, once daily (QD) until achievement of major molecular response (MMR) up to 12 months. Once MMR was achieved, participants received reduced dose of ponatinib 15 mg orally once daily up to approximately 42 months.
- Cohort B: Ponatinib 15 mg: Ponatinib 15 mg, tablets, orally, QD until achievement of MMR up to 12 months. Once MMR was achieved, participants received reduced dose of ponatinib 15 mg orally once daily up to approximately 45 months.
Period: Overall Study
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Started | 11 | 21 | 12
Completed | 0 | 0 | 0
Not Completed | 11 | 21 | 12
Not completed — Adverse event (not progressive disease) | 1 | 4 | 1
Not completed — Progressive disease | 1 | 3 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 5 | 10 | 6
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Reason not Specified | 0 | 0 | 1
Not completed — Randomized but not Treated | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who have received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg | Total
Number analyzed (Participants) | 10 | 21 | 12 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (17.43) | 44.7 (15.53) | 54.3 (13.23) | 47.16 (15.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 6 | 20
  Male | 7 | 10 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 21 | 11 | 42
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 16 | 10 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 0 | 1 | 0 | 1
  Canada | 0 | 0 | 1 | 1
  Czech Republic | 0 | 0 | 2 | 2
  France | 1 | 1 | 1 | 3
  Hungary | 0 | 1 | 0 | 1
  Italy | 0 | 0 | 1 | 1
  Korea, North | 1 | 2 | 0 | 3
  Russia | 8 | 16 | 7 | 31
Height [Mean (Standard Deviation); unit: cm] — Population: Number analyzed is the number of participants with data available for Height at Baseline.
  cm
    number analyzed (Participants) | 10 | 21 | 11 | 42
    (all) | 172.9 (9.62) | 169.4 (9.35) | 168.8 (9.17) | 170.1 (9.28)
Weight [Mean (Standard Deviation); unit: kg] | 77.50 (18.335) | 72.72 (15.213) | 70.94 (14.711) | 73.34 (15.65)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI is calculated as weight (kg) divided by square of height (m^2). Population: Number analyzed is the number of participants with data available for BMI at Baseline.
  kg/m^2
    number analyzed (Participants) | 10 | 21 | 11 | 42
    (all) | 25.90 (5.870) | 25.35 (4.974) | 25.18 (4.442) | 25.44 (4.95)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Molecular Response (MMR)
Description: MMR is defined as the percentage of participants achieving a ratio of ≤0.1% Breakpoint Cluster Region-Abelson (BCR ABL) to ABL transcripts on the international scale (≤0.1% BCR-ABL/ABL[IS]) at any time within 12 months after randomization.
Time Frame: Up to 12 months
Population: Safety Population included all participants who have received at least 1 dose of study drug, with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 11
percentage of participants | 50.0 [18.7 to 81.3] | 33.3 [14.6 to 57.0] | 45.5 [16.7 to 76.6]

2. Secondary Outcome: Percentage of Participants With Major Cytogenetic Response (MCyR)
Description: MCyR was the percentage of participants achieving Complete cytogenetic response (CCyR: defined as 0% Philadelphia chromosome-positive [Ph+] metaphases by cytogenetic analysis of bone marrow) or Partial Cytogenetic Response (PCyR: defined as >0% to 35% Ph+ metaphases by cytogenetic analysis of bone marrow) at any time within 12 months after randomization.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 20 | 12
percentage of participants | 50.0 [18.7 to 81.3] | 60.0 [36.1 to 80.9] | 50.0 [21.1 to 78.9]

3. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR)
Description: CCyR rate was defined as the percentage of participants achieving CCyR up to 12 months after randomization. CCyR is defined as 0% Philadelphia chromosome-positive [Ph+] metaphases by cytogenetic analysis of bone marrow.
Time Frame: Up to 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 20 | 12
percentage of participants | 40.0 [12.2 to 73.8] | 55.0 [31.5 to 76.9] | 50.0 [21.1 to 78.9]

4. Secondary Outcome: Percentage of Participants With Molecular Response (MR)
Description: Molecular response rate is defined as percentage of participants achieving MR2: Molecular response with 2-log reduction (defined as ≤1% BCR-ABL[IS]), MMR: Major molecular responder, MR4 (defined as ≤0.01% BCR-ABL[IS]), and MR4.5 (defined as ≤0.0032% BCR-ABL[IS]) after randomization.
Time Frame: From Month 3 to every 3 months up to 48 months
Population: Safety Population included all participants who have received at least 1 dose of study drug, with data available for analysis. Number analyzed are participants with data available for analyses at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 12
percentage of participants
  MR2 - Month 3: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 3 | 70.0 | 38.1 | 45.5
  MR2 - Month 6: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 6 | 60.0 | 57.1 | 54.5
  MR2 - Month 9: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 9 | 50.0 | 52.4 | 45.5
  MR2 - Month 12: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 12 | 50.0 | 52.4 | 54.5
  MR2 - Month 15: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 15 | 50.0 | 52.4 | 54.5
  MR2 - Month 18: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 18 | 50.0 | 47.6 | 54.5
  MR2 - Month 21: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 21 | 50.0 | 52.4 | 45.5
  MR2 - Month 24: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 24 | 50.0 | 47.6 | 54.5
  MR2 - Month 27: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 27 | 50.0 | 42.9 | 54.5
  MR2 - Month 30: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 30 | 50.0 | 38.1 | 45.5
  MR2 - Month 33: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 33 | 30.0 | 33.3 | 27.3
  MR2 - Month 36: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 36 | 50.0 | 33.3 | 36.4
  MR2 - Month 39: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 39 | 20.0 | 14.3 | 18.2
  MR2 - Month 42: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 42 | 10.0 | 9.5 | 9.1
  MR2 - Month 45: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 45 | 10.0 | 14.3 | 9.1
  MR2 - Month 48: number analyzed (Participants) | 10 | 21 | 11
  MR2 - Month 48 | 10.0 | 4.8 | 9.1
  MR3/MMR - Month 3: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 3 | 30.0 | 4.8 | 18.2
  MR3/MMR - Month 6: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 6 | 30.0 | 28.6 | 36.4
  MR3/MMR - Month 9: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 9 | 30.0 | 28.6 | 45.5
  MR3/MMR - Month 12: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 12 | 40.0 | 33.3 | 45.5
  MR3/MMR - Month 15: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 15 | 40.0 | 28.6 | 45.5
  MR3/MMR - Month 18: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 18 | 40.0 | 38.1 | 45.5
  MR3/MMR - Month 21: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 21 | 40.0 | 33.3 | 45.5
  MR3/MMR - Month 24: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 24 | 40.0 | 33.3 | 45.5
  MR3/MMR - Month 27: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 27 | 40.0 | 33.3 | 45.5
  MR3/MMR - Month 30: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 30 | 40.0 | 33.3 | 45.5
  MR3/MMR - Month 33: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 33 | 20.0 | 28.6 | 27.3
  MR3/MMR - Month 36: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 36 | 40.0 | 28.6 | 36.4
  MR3/MMR - Month 39: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 39 | 20.0 | 14.3 | 18.2
  MR3/MMR - Month 42: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 42 | 10.0 | 9.5 | 9.1
  MR3/MMR - Month 45: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 45 | 10.0 | 9.5 | 9.1
  MR3/MMR - Month 48: number analyzed (Participants) | 10 | 21 | 11
  MR3/MMR - Month 48 | 10.0 | 4.8 | 9.1
  MR4 - Month 3: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 3 | 0.0 | 0.0 | 0.0
  MR4 - Month 6: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 6 | 20.0 | 14.3 | 9.1
  MR4 - Month 9: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 9 | 10.0 | 9.5 | 18.2
  MR4 - Month 12: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 12 | 10.0 | 9.5 | 27.3
  MR4 - Month 15: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 15 | 10.0 | 19.0 | 27.3
  MR4 - Month 18: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 18 | 20.0 | 23.8 | 27.3
  MR4 - Month 21: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 21 | 20.0 | 9.5 | 36.4
  MR4 - Month 24: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 24 | 10.0 | 19.0 | 36.4
  MR4 - Month 27: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 27 | 20.0 | 19.0 | 36.4
  MR4 - Month 30: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 30 | 20.0 | 14.3 | 36.4
  MR4 - Month 33: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 33 | 0.0 | 14.3 | 9.1
  MR4 - Month 36: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 36 | 10.0 | 19.0 | 27.3
  MR4 - Month 39: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 39 | 20.0 | 4.8 | 18.2
  MR4 - Month 42: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 42 | 10.0 | 0.0 | 9.1
  MR4 - Month 45: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 45 | 10.0 | 4.8 | 9.1
  MR4 - Month 48: number analyzed (Participants) | 10 | 21 | 11
  MR4 - Month 48 | 10.0 | 0.0 | 9.1
  MR4.5 - Month 3: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 3 | 0.0 | 0.0 | 0.0
  MR4.5 - Month 6: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 6 | 20.0 | 0.0 | 0.0
  MR4.5 - Month 9: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 9 | 0.0 | 4.8 | 9.1
  MR4.5 - Month 12: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 12 | 0.0 | 4.8 | 18.2
  MR4.5 - Month 15: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 15 | 10.0 | 4.8 | 9.1
  MR4.5 - Month 18: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 18 | 10.0 | 9.5 | 9.1
  MR4.5 - Month 21: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 21 | 10.0 | 9.5 | 27.3
  MR4.5 - Month 24: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 24 | 10.0 | 4.8 | 18.2
  MR4.5 - Month 27: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 27 | 10.0 | 14.3 | 18.2
  MR4.5 - Month 30: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 30 | 10.0 | 4.8 | 27.3
  MR4.5 - Month 33: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 33 | 0.0 | 4.8 | 0.0
  MR4.5 - Month 36: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 36 | 10.0 | 9.5 | 18.2
  MR4.5 - Month 39: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 39 | 10.0 | 4.8 | 18.2
  MR4.5 - Month 42: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 42 | 10.0 | 0.0 | 9.1
  MR4.5 - Month 45: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 45 | 10.0 | 0.0 | 9.1
  MR4.5 - Month 48: number analyzed (Participants) | 10 | 21 | 11
  MR4.5 - Month 48 | 0.0 | 0.0 | 9.1

5. Secondary Outcome: Percentage of Participants With MR1
Description: MR1 was defined as the percentage of participants achieving a ratio of ≤10% BCR ABL to ABL transcripts on the international scale at 3 months.
Time Frame: Month 3
Population: Safety Population includes all participants who have received at least 1 dose of study drug, with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 11
percentage of participants | 70.0 | 66.7 | 63.6

6. Secondary Outcome: Percentage of Participants With Treatment Emergent Arterial Occlusive Events (TE-AOEs), Treatment Emergent Venous Thromboembolic Events (TE-VTE), Adverse Events (AEs), and Serious AEs (SAEs)
Description: TE-AOE: arterial occlusive event with an initial onset date on or after first dose date and no later than 30 days after last dose date of study treatment or events starting after initial consent that worsen in severity on or after first dose date. TE-VTE: vascular occlusive event with an initial onset date on or after first dose date and no later than 30 days after last dose date of study treatment or events starting after initial consent that worsen in severity on or after first dose date. AE: any untoward medical occurrence in participant administered pharmaceutical product; untoward medical occurrence does not necessarily have causal relationship with this treatment. SAE: any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is congenital anomaly/birth defect/is medically important event.
Time Frame: From first dose up to 30 days post last dose (Up to approximately 46 months)
Population: Safety Population includes all participants who have received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 12
percentage of participants
  TE-AOE | 0 | 4.8 | 8.3
  TE-VOEs | 0 | 0 | 0
  AEs | 100 | 95.2 | 100
  SAEs | 40.0 | 14.3 | 16.7

7. Secondary Outcome: Time to Response
Description: Time to MMR defined as the interval between the randomization date and the first date at which the criteria for response was met. MMR was defined as <=0.1% BCR-ABL.
Time Frame: Up to approximately 60 months
Population: Safety Population includes all participants who have received at least 1 dose of study drug. Only responders were analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 5 | 9 | 5
months | 3.07 [3.0 to NA] — The upper limit of confidence interval (CI) was not estimable due to less number of participants with event. | 6.29 [3.0 to 18.1] | 6.07 [3.0 to NA] — The upper limit of CI was not estimable due to less number of participants with event.

8. Secondary Outcome: Duration of Response
Description: Duration of response defined as the interval between the first assessment at which the criteria for response was met until the earliest date at which loss of response occurs, or the criteria for progression was met.
Time Frame: Up to approximately 60 months
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 5 | 9 | 5
months | NA [NA to NA] — The median, lower limit and upper limit of CI were not estimable due to less number of participants with event. | NA [3.0 to NA] — The median and upper limit of CI were not estimable due to less number of participants with event. | NA [NA to NA] — The median, lower limit and upper limit of CI were not estimable due to less number of participants with event.

9. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) defined as the interval between the first dose date of study treatment and the first date at which the criteria for progression was met (progression to AP- or BP CML), or death due to any cause, censored at the last response assessment.
Time Frame: Up to end of study (approximately 60 months)
Population: Safety Population includes all participants who have received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 12
months | NA [8.0 to NA] — The median and upper limit of CI were not estimable due to less number of participants with event. | NA [NA to NA] — The median, lower limit and upper limit of CI were not estimable due to less number of participants with event. | NA [NA to NA] — The median, lower limit and upper limit of CI were not estimable due to less number of participants with event.

10. Secondary Outcome: Overall Survival
Description: Overall survival (OS) defined as the interval between the first dose date of study treatment and date of death due to any cause, censored at the last contact date to be alive.
Time Frame: Up to end of study (approximately 60 months)
Population: Safety Population includes all participants who have received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort B: Ponatinib 15 mg: Ponatinib 15 mg, tablets, orally, QD until achievement of MMR up to 12 months. Once MMR was achieved, participants received reduced dose of ponatinib 15 mg orally once daily up to approximately 45months.
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 12
months | NA [18.5 to NA] — The median and upper limit of CI were not estimable due to less number of participants with event. | NA [NA to NA] — The median, lower limit and upper limit of CI were not estimable due to less number of participants with event. | NA [NA to NA] — The median, lower limit and upper limit of CI were not estimable due to less number of participants with event.

11. Secondary Outcome: Percentage of Participants Who Achieved/Maintained Complete Hematologic Response (CHR)
Description: CHR rate is defined as the percentage of participants achieving CHR at any time after initiation of study treatment. CHR is defined as achieving all of the following measurements: White blood cells (WBC) ≤ institutional upper limit of normal (ULN); Platelets <450 x 10^9/L; No blasts or promyelocytes in peripheral blood; <5% myelocytes plus metamyelocytes in peripheral blood; Basophils in peripheral blood <5%; No extramedullary involvement (including no hepatomegaly or splenomegaly).
Time Frame: 3 months after the first dose of study treatment
Population: Safety Population includes all participants who have received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 12
percentage of participants | 60.0 [26.2 to 87.8] | 81.0 [58.1 to 94.6] | 50.0 [21.1 to 78.9]

12. Secondary Outcome: Percentage of Participants With Treatment Emergent AEs Leading to Treatment Discontinuation, Dose Reduction and Dose Interruption
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose up to end of treatment (Up to approximately 45 months)
Population: Safety Population includes all participants who have received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 10 | 21 | 12
percentage of participants
  TEAEs Leading to Treatment Discontinuation | 10.0 | 23.8 | 25.0
  TEAEs Leading to Dose Reduction | 40.0 | 19.0 | 33.3
  TEAEs Leading to Dose Interruption | 70.0 | 38.1 | 41.7

13. Secondary Outcome: Percentage of Participants With Progression to Accelerated Phase (AP) or Blast Phase (BP)-CML
Description: Progression to AP is defined as: >=15% and <30% blasts in peripheral blood or bone marrow or >=20% basophils in peripheral blood or bone marrow or >=30% blasts + promyelocytes in peripheral blood or bone marrow (but <30% blasts) or <100*10^9 platelets/L in peripheral blood unrelated to therapy or cytogenetic, genetic evidence of clonal evolution, and no extramedullary disease. Progression to BP-CML is defined as: >=30% blasts in peripheral blood or bone marrow or extramedullary disease other than hepatosplenomegaly.
Time Frame: Up to end of study (Up to approximately 60 months)
Population: As the study was terminated, data was not collected and analyzed for this outcome measure.
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From first dose up to end of study (Up to approximately 60 months); for serious and other adverse events: from first dose up to 30 days post last dose (Up to approximately 46 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Population includes all participants who have received at least 1 dose of study drug.
Arm/Group | Cohort A: Ponatinib 30 mg | Cohort B: Ponatinib 15 mg | Cohort C: Nilotinib 400 mg
All-Cause Mortality (participants affected / at risk) | 1/10 | 1/21 | 0/12
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/21 | 2/12
Other Adverse Events (participants affected / at risk) | 10/10 | 20/21 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ponatinib 30 mg (N=10) | Cohort B: Ponatinib 15 mg (N=21) | Cohort C: Nilotinib 400 mg (N=12)
Pneumonia (Infections and infestations) | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ponatinib 30 mg (N=10) | Cohort B: Ponatinib 15 mg (N=21) | Cohort C: Nilotinib 400 mg (N=12)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 5 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 2
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 3 | 1 | 2
Blood cholesterol increased (Investigations) | 2 | 2 | 3
Platelet count decreased (Investigations) | 2 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2
Lipase increased (Investigations) | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 0
Platelet count increased (Investigations) | 1 | 1 | 0
Weight increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Hypertriglyceridaemia (Gastrointestinal disorders) | 1 | 2 | 0
Hyperglycaemia (Gastrointestinal disorders) | 1 | 1 | 0
Diabetes mellitus (Gastrointestinal disorders) | 1 | 0 | 0
Hyperlipidaemia (Gastrointestinal disorders) | 1 | 0 | 0
Hypophosphataemia (Gastrointestinal disorders) | 0 | 1 | 1
Hypophosphataemia (Gastrointestinal disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Paternal exposure timing unspecified (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 2 | 1
Essential hypertension (Vascular disorders) | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Dilatation atrial (Cardiac disorders) | 0 | 0 | 1
Right atrial hypertrophy (Cardiac disorders) | 0 | 0 | 1
Right ventricular dilatation (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1
Retinal vascular disorder (Eye disorders) | 1 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 3
Pyrexia (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary artery dilatation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Ocular icterus (Hepatobiliary disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
This study was terminated due to operational feasibility and not due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02627677/Prot_000.pdf
  • Statistical Analysis Plan (2016-07-31): https://cdn.clinicaltrials.gov/large-docs/77/NCT02627677/SAP_001.pdf